CLINICAL TRIAL: NCT00370331
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study, to Evaluate the Efficacy, Safety and Tolerability of Eltrombopag Olamine (SB-497115-GR), a Thrombopoietin Receptor Agonist, Administered for 6 Months as Oral Tablets Once Daily in Adult Subjects With Previously Treated Chronic ITP.
Brief Title: RAISE: Randomized Placebo-Controlled Idiopathic Thrombocytopenic Purpura (ITP) Study With Eltrombopag
Acronym: RAISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRA102537
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: ITP; idiopathic; platelets; purpura; thrombocytopenia; Idiopathic Thrombocytopenic Purpura; thrombocytopenic
MeSH Terms: conditions — Purpura; Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment arm plus standard of care (Experimental): Subjects will initiate treatment with 50 mg eltrombopag or matching placebo once daily. Based upon the subjects platelet count at each visit, the dose of eltrombopag may be adjusted either up or down.
  Interventions: Drug: eltrombopag
- placebo plus standard of care (Placebo Comparator): Subjects will initiate treatment with 50 mg eltrombopag or matching placebo once daily. Based upon the subjects platelet count at each visit, the dose of eltrombopag may be adjusted either up or down.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eltrombopag — Subjects will initiate treatment with either 50 mg eltrombopag or matching placebo once daily. Based upon the subjects platelet count at each visit, the dose of eltrombopag may be adjusted either up or down.
  Arms: Treatment arm plus standard of care
Drug: Placebo — Subjects will initiate treatment with either 50 mg eltrombopag or matching placebo once daily. Based upon the subjects platelet count at each visit, the dose of eltrombopag may be adjusted either up or down
  Arms: placebo plus standard of care

SUMMARY:
The rationale for this Phase III study is to evaluate the 6 month safety and efficacy of eltrombopag in the treatment of previously treated subjects with chronic ITP. The starting dose of eltrombopag, 50 mg, once daily was selected based upon the observed efficacy, safety and pharmacokinetics in a dose-finding Study (TRA100773). This Phase III study is a randomized, double-blind, placebo-controlled, Phase III study, to evaluate efficacy, safety and tolerability of eltrombopag, initially administered as 50 mg oral tablets once daily for six months in adult subjects with previously treated chronic ITP. Subjects will be randomized 2:1, eltrombopag to placebo, and will be stratified based upon splenectomy status, use of ITP medication at baseline and baseline platelet count less than or equal to 15,000/µL. Subjects will receive study medication for 6 months, during which the dose of study medication may be adjusted based upon individual platelet counts. In addition, subjects may taper off concomitant ITP medications and may receive any rescue treatments as dictated by local standard of care. After discontinuation of study medication, subjects will complete follow-up visits at weeks 1, 2, 4 and months 3 and 6.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled phase III study, to evaluate the efficacy, safety and tolerability of eltrombopag olamine (SB-497115-GR), a thrombopoietin receptor agonist, administered for 6 months as oral tablets once daily in adult subjects with previously treated chronic idiopathic thrombocytopenic purpura (ITP).

ELIGIBILITY:
Inclusion criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Subject has signed and dated a written informed consent.
* Adults (≥18 years) diagnosed with chronic ITP according to the American Society for Hematology/British Committee for Standards in Hematology (ASH/BCSH) guidelines [George, 1996; BCSH, 2003], and platelet count < 30,000/μL on Day 1 (or within 24 hours prior to dosing on Day 1). In addition, a peripheral blood smear should support the diagnosis of ITP with no evidence of other causes of thrombocytopenia (e.g. pseudothrombocytopenia, myelofibrosis). The physical examination should not suggest any disease which may cause thrombocytopenia other than ITP.
* Subjects who have previously received one or more prior ITP therapies. Previous treatments for ITP include but are not limited to corticosteroids, immunoglobulins, azathioprine, danazol, cyclophosphamide and/or rituximab.
* Subjects must have either initially responded (platelet count > 100,000/μL) to a previous ITP therapy or have had a bone marrow examination consistent with ITP within 3 years to rule out myelodysplastic syndromes or other causes of thrombocytopenia.
* Previous therapy for ITP with immunoglobulins (IVIg and anti-D) must have been completed at least 1 week prior to randomization and the platelet count must show a clear downward trend after the last treatment with immunoglobulins. Previous treatment for ITP with splenectomy, rituximab and cyclophosphamide must have been completed at least 4 weeks prior to randomization, or clearly be ineffective.
* Subjects treated with concomitant ITP medication (e.g. corticosteroids or azathioprine) must be receiving a dose that has been stable for at least 4 weeks prior to randomization. Subjects treated with cyclosporine A, mycophenolate mofetil or danazol must be receiving a dose that has been stable for at least 3 months prior to randomization. The medication should be continued with a stable dose for the initial 6 weeks of study "Concomitant ITP Therapy")
* Prothrombin time (PT/INR) and activated partial thromboplastin time (aPTT) must be within 80 to 120% of the normal range with no history of hypercoagulable state.
* A complete blood count (CBC), within the reference range (including WBC differential not indicative of a disorder other than ITP), with the following exceptions:
* < 30,000 platelets/μL on Day 1 (or within 24 hours of Day 1) is required for inclusion,
* Hemoglobin: Subjects with hemoglobin levels between 10 g/dL (100 g/L) and the lower limit of normal are eligible for inclusion, if anemia is clearly attributable to ITP (excessive blood loss).
* ANC ≥ 1500/μL (1.5 x 10^9/L) is required for inclusion (elevated WBC/ANC due to steroid treatment is acceptable).
* The following clinical chemistries MUST NOT exceed the upper limit of normal (ULN) reference range by more than 20%: creatinine, ALT, AST, total bilirubin, and alkaline phosphatase. In addition, total albumin must not be below the lower limit of normal (LLN) by more than 10%.
* Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use one of the following highly effective methods of contraception (i.e., Pearl Index <1.0%) from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:
* Complete abstinence from intercourse;
* Intrauterine device (IUD);
* Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide);
* Male partner is sterile prior to entry into the study and is the only partner of the female;
* Systemic contraceptives (combined or progesterone only). Subject is able to understand and comply with protocol requirements and instructions and intends to complete the study as planned.

Exclusion criteria:

* A subject will NOT be eligible for inclusion in this study if any of the following criteria apply:
* Any clinically relevant abnormality, other than ITP, identified on the screening examination or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another primary diagnosis (e.g., thrombocytopenia is secondary to another disease).
* Concurrent malignant disease and/or history of cancer treatment with cytotoxic chemotherapy and/or radiotherapy.
* Any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, etc), or any other family history of arterial or venous thrombosis.
* Pre-existing cardiovascular disease (congestive heart failure, New York Heart Association [NYHA] Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec.
* Female subjects who are nursing or pregnant (positive serum or urine b-human chorionic gonadotrophin pregnancy test) at screening or pre-dose on Day 1.
* History of alcohol/drug abuse.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* Subject treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDs) or anti-coagulants for > 3 consecutive days within 2 weeks of the study start and until the end of the study.
* History of platelet agglutination abnormality that prevents reliable measurement of platelet counts.
* All subjects with secondary immune thrombocytopenia, including those with laboratory or clinical evidence of HIV infection, anti-phospholipid antibody syndrome, chronic hepatitis B infection, hepatitis C virus infection, or any evidence for active hepatitis at the time of subject screening. If a potential subject has no clinical history that would support HIV infection or hepatitis infection, no further laboratory screening is necessary; however, standard medical practice would suggest further evaluation of patients who have risk factors for these infections.
* Previous participation in a clinical study with eltrombopag.
* Patients planning to have cataract surgery.
* In France, a subject is neither affiliated with nor a beneficiary of a social security category.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (101):
- United States (23):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Lawton, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Willow Grove, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
- GSK Investigational Site, Vienna, Austria
- Canada (7):
  - GSK Investigational Site, Burnaby, British Columbia
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Weston, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
- China (3):
  - GSK Investigational Site, Jiang Su Province
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
- GSK Investigational Site, Odense, Denmark
- GSK Investigational Site, Kuopio, Finland
- France (4):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Pessac
- Germany (5):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Saarbrücken, Saarland
  - GSK Investigational Site, Berlin, State of Berlin
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Shatin, Hong Kong
- India (2):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Manipal
- Italy (6):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Albano Laziale (Roma), Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Padua, Veneto
  - GSK Investigational Site, Vicenza, Veneto
- Netherlands (3):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Zwolle
- New Zealand (3):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Grafton
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Lima
- Poland (7):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Legnica
  - GSK Investigational Site, Opole
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Wroclaw
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
- Slovakia (3):
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Prešov
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
- GSK Investigational Site, Taipei, Taiwan
- Tunisia (3):
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Sousse
  - GSK Investigational Site, Tunis
- Ukraine (4):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Odesa
- United Kingdom (8):
  - GSK Investigational Site, Plymouth, Devon
  - GSK Investigational Site, Taunton, Somerset
  - GSK Investigational Site, Leed
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Morriston
  - GSK Investigational Site, Reading
  - GSK Investigational Site, Rhyl, Denbighshire
- GSK Investigational Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Cheng G, Saleh MN, Marcher C, Vasey S, Mayer B, Aivado M, Arning M, Stone NL, Bussel JB. Eltrombopag for management of chronic immune thrombocytopenia (RAISE): a 6-month, randomised, phase 3 study. Lancet. 2011 Jan 29;377(9763):393-402. doi: 10.1016/S0140-6736(10)60959-2. Epub 2010 Aug 23. PMID 20739054
- [Background] Haselboeck J, Pabinger I, Ay C, Koder S, Panzer S. Platelet activation and function during eltrombopag treatment in immune thrombocytopenia. Ann Hematol. 2012 Jan;91(1):109-13. doi: 10.1007/s00277-011-1249-5. Epub 2011 May 7. PMID 21553010
- [Background] Hayes S, Ouellet D, Zhang J, Wire MB, Gibiansky E. Population PK/PD modeling of eltrombopag in healthy volunteers and patients with immune thrombocytopenic purpura and optimization of response-guided dosing. J Clin Pharmacol. 2011 Oct;51(10):1403-17. doi: 10.1177/0091270010383019. Epub 2010 Dec 8. PMID 21148042
- [Background] Tarantino MD, Fogarty P, Mayer B, Vasey SY, Brainsky A. Efficacy of eltrombopag in management of bleeding symptoms associated with chronic immune thrombocytopenia. Blood Coagul Fibrinolysis. 2013 Apr;24(3):284-96. doi: 10.1097/MBC.0b013e32835fac99. PMID 23492914
- [Derived] Fogarty PF, Tarantino MD, Brainsky A, Signorovitch J, Grotzinger KM. Selective validation of the WHO Bleeding Scale in patients with chronic immune thrombocytopenia. Curr Med Res Opin. 2012 Jan;28(1):79-87. doi: 10.1185/03007995.2011.644849. Epub 2011 Dec 20. PMID 22117897
- [Derived] Signorovitch J, Brainsky A, Grotzinger KM. Validation of the FACIT-fatigue subscale, selected items from FACT-thrombocytopenia, and the SF-36v2 in patients with chronic immune thrombocytopenia. Qual Life Res. 2011 Dec;20(10):1737-44. doi: 10.1007/s11136-011-9912-9. Epub 2011 May 1. PMID 21533818

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo tablets taken once a day
- Eltrombopag 50 mg QD: Eltrombopag 50 mg oral tablets taken once a day (QD)
Period: Overall Study
Arm/Group | Placebo | Eltrombopag 50 mg QD
Started | 62 | 135
Completed | 55 | 112
Not Completed | 7 | 23
Not completed — Adverse Event | 4 | 13
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 0 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Non-compliance | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Eltrombopag 50 mg QD | Total
Number analyzed (Participants) | 62 | 135 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (14.72) | 46.5 (15.61) | 47.9 (15.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 93 | 136
  Male | 19 | 42 | 61
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African | 1 | 2 | 3
  American Indian/Alaska native | 4 | 8 | 12
  East Asian | 10 | 19 | 29
  South-East Asian | 3 | 2 | 5
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White/Arabic/North African | 2 | 6 | 8
  White/Caucasian/European | 42 | 95 | 137
  Mixed Race | 0 | 2 | 2
Stratification variable [Number; unit: Participants] — Subjects were stratified at randomization based on current use of idiopathic thrombocytopenic purpura (ITP) medication, splenectomy status, and baseline platelet count
  Participants
    Use of ITP medication at randomization | 31 | 63 | 94
    Splenectomy at randomization | 21 | 50 | 71
    Platelet count less or equal 15,000 per microliter | 30 | 67 | 97

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders
Description: The percentage of evaluable participants who achieved a platelet response (defined as a platelet count between 50,000 and 400,000 microliter) at each nominal on-therapy day and 4 weeks post-treatment
Time Frame: Baseline; each on-therapy treatment day; Weeks 10, 14, 18, 22, and 26; and Weeks 1, 2, and 4 post-treatment
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Percentage of participants
  Baseline | 2 | 1
  Day 8 | 7 | 37
  Day 15 | 8 | 46
  Day 22 | 8 | 51
  Day 29 | 10 | 49
  Day 36 | 8 | 56
  Day 43 | 14 | 54
  Week 10 | 17 | 52
  Week 14 | 18 | 46
  Week 18 | 17 | 46
  Week 22 | 19 | 49
  Week 26 | 17 | 52
  1 Week Follow-up | 15 | 42
  2 Week Follow-up | 18 | 22
  4 Week Follow-up | 14 | 20
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 50 mg QD; Test type: Superiority or Other; p < 0.001, Repeated measures model for binary data; Repeated measures model for binary data using Generalized Estimating Equations (GEE); Odds Ratio (OR) = 8.2, 99% CI [3.59 to 18.73]

2. Secondary Outcome: Summary of Median Platelet Counts
Description: Platelet counts were measured by blood draw.
Time Frame: Baseline; Day 8 through Week 26 on-treatment; and 1, 2, 4 week follow-up visits
Population: ITT Population
Measure: Median (Full Range); unit: platelets/microliter (ul)
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
platelets/microliter (ul)
  Baseline | 16,000 [2000 to 87,000] | 16,000 [0 to 78,000]
  Day 8 | 17,500 [3000 to 354,000] | 36,000 [1000 to 593,000]
  Day 15 | 18,000 [2000 to 214,000] | 54,000 [2000 to 750,000]
  Day 22 | 18,500 [1000 to 271,000] | 54,000 [1000 to 507,000]
  Day 29 | 18,000 [3000 to 313,000] | 53,000 [1000 to 400,000]
  Day 36 | 19,000 [4000 to 297,000] | 60,000 [1000 to 952,000]
  Day 43 | 20,000 [3000 to 275,000] | 59,000 [1000 to 545,000]
  Week 10 | 20,000 [0 to 293,000] | 61,500 [1000 to 433,000]
  Week 14 | 17,500 [1000 to 303,000] | 60,000 [1000 to 409,000]
  Week 18 | 20,500 [2000 to 281,000] | 61,000 [3000 to 363,000]
  Week 22 | 23,000 [1000 to 315,000] | 72,000 [3000 to 408,000]
  Week 26 | 23,000 [2000 to 315,000] | 73,500 [1000 to 429,000]
  1 Week Follow-up | 19,000 [0 to 323,000] | 38,500 [1000 to 409,000]
  2 Week Follow-up | 18,000 [1000 to 340,000] | 21,000 [1000 to 434,000]
  4 Week Follow-up | 18,000 [1000 to 301,000] | 24,000 [1000 to 446,000]

3. Secondary Outcome: Percentage of Participants Initiating Rescue Treatment On-therapy
Description: Percentage of participants initiating new ITP medication, an increased dose of concomitant ITP medication from baseline, platelet transfusion, or splenectomy.
Time Frame: Anytime from Day 1 to Week 26
Population: All participants randomized to receive placebo or eltrombopag treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Percentage of participants
  Participants who received rescue treatment | 40 | 18
  Participants who did not receive rescue treatment | 60 | 82

4. Secondary Outcome: Maximum and Total Weeks of Platelet Response
Description: Response is defined as a platelet count between 50,000 and 400,000 platelets per microliter.
Time Frame: Day 1 through Week 26 on-treatment
Population: ITT Population
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Weeks
  Maximum continuous Response | 0 [0 to 25] | 8.1 [0 to 26]
  Cumulative Response | 0 [0 to 25] | 10.9 [0 to 26]

5. Secondary Outcome: Percentage of Participants With a Reduction in Use of Baseline ITP Medication
Description: Percentage of participants who experienced a reduction in their baseline concomitant ITP medication use
Time Frame: From Day 1 through Week 26 on-treatment
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 60 | 134
Percentage of participants
  Participants who reduced/discontinued ITP therapy | 32 | 59
  Participants not reducing/discont. ITP therapy | 68 | 41

6. Secondary Outcome: WHO Bleeding Scale
Description: Summary of World Health Organization (WHO) bleeding scores at each nominal visit. WHO Grades 1-4 = any bleeding; WHO Grades 2-4 = clinically significant bleeding
Time Frame: Baseline, all nominal visits on-therapy defined as Day 8, Day 15, Day 22, Day 29, Day 36, Day 43, Week 10, Week 14, Week 18, Week 22, Week 26, and 1, 2 and 4 week follow-up visits
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Percentage of participants
  Baseline, WHO Grades 1-4 | 77 | 73
  Day 8, WHO Grades 1-4 | 73 | 56
  Day 15, WHO Grades 1-4 | 68 | 39
  Day 22, WHO Grades 1-4 | 67 | 38
  Day 29, WHO Grades 1-4 | 56 | 37
  Day 36, WHO Grades 1-4 | 66 | 23
  Day 43, WHO Grades 1-4 | 59 | 23
  Week 10, WHO Grades 1-4 | 49 | 22
  Week 14, WHO Grades 1-4 | 57 | 23
  Week 18, WHO Grades 1-4 | 59 | 22
  Week 22, WHO Grades 1-4 | 46 | 18
  Week 26, WHO Grades 1-4 | 56 | 22
  1 Week Follow-up, WHO Grades 1-4 | 59 | 28
  2 Week Follow-up, WHO Grades 1-4 | 56 | 50
  4 Week Follow-up, WHO Grades 1-4 | 59 | 46
  Baseline, WHO Grades 2-4 | 28 | 22
  Day 8, WHO Grades 2-4 | 20 | 16
  Day 15, WHO Grades 2-4 | 22 | 8
  Day 22, WHO Grades 2-4 | 21 | 11
  Day 29, WHO Grades 2-4 | 19 | 10
  Day 36, WHO Grades 2-4 | 19 | 7
  Day 43, WHO Grades 2-4 | 19 | 5
  Week 10, WHO Grades 2-4 | 13 | 9
  Week 14, WHO Grades 2-4 | 17 | 5
  Week 18, WHO Grades 2-4 | 18 | 2
  Week 22, WHO Grades 2-4 | 10 | 8
  Week 26, WHO Grades 2-4 | 15 | 7
  1 Week Follow-up, WHO Grades 2-4 | 20 | 11
  2 Week Follow-up, WHO Grades 2-4 | 18 | 16
  4 Week Follow-up, WHO Grades 2-4 | 21 | 13

7. Secondary Outcome: HR-QoL Instrument and Domain Scores From the SF-36v2 Questionnaire at Baseline, Week 6, Week 14, and Week 26 or Early Discontinuation From Study Treatment
Description: Health-related quality of life (HR-QoL) patient reported outcomes from the short form-36v2 (SF-36v2) questionnaire. Scores could range from 0 (worst possible) to 100 (best possible).
Time Frame: Baseline, Week 6, Week 14, and Week 26/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Points on a scale (0-100)
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Points on a scale (0-100)
  SF-36v2 physical function, Baseline | 75.0 (21.7) | 73.1 (26.8)
  SF-36v2 physical function, Week 6 | 76.5 (20.8) | 78.0 (24.4)
  SF-36v2 physical function, Week 14 | 77.6 (20.0) | 78.9 (22.5)
  SF-36v2 physical funct., Week 26/Early Withdrawal | 75.8 (22.6) | 80.6 (21.7)
  SF-36v2 physical role, Baseline | 64.5 (26.7) | 64.5 (30.5)
  SF-36v2 physical role, Week 6 | 66.9 (25.4) | 73.7 (27.4)
  SF-36v2 physical role, Week 14 | 67.2 (25.8) | 72.9 (24.9)
  SF-36v2 physical role, Week 26/Early Withdrawal | 67.5 (27.1) | 73.7 (25.4)
  SF-36v2 bodily pain, Baseline | 70.0 (23.2) | 75.2 (27.8)
  SF-36v2 bodily pain, Week 6 | 69.9 (25.9) | 78.5 (25.4)
  SF-36v2 bodily pain, Week 14 | 68.3 (24.8) | 77.6 (25.8)
  SF-36v2 bodily pain, Week 26/Early Withdrawal | 68.5 (25.0) | 75.7 (26.6)
  SF-36v2 general health, Baseline | 53.7 (21.8) | 56.0 (21.3)
  SF-36v2 general health, Week 6 | 55.9 (21.4) | 59.7 (21.5)
  SF-36v2 general health, Week 14 | 52.8 (23.2) | 59.3 (20.7)
  SF-36v2 general health, Week 26/Early Withdrawal | 53.3 (24.9) | 57.3 (23.1)
  SF-36v2 vitality, Baseline | 56.7 (20.2) | 55.1 (26.3)
  SF-36v2 vitality, Week 6 | 59.0 (20.0) | 62.1 (22.7)
  SF-36v2 vitality, Week 14 | 56.8 (22.3) | 61.0 (22.4)
  SF-36v2 vitality, Week 26/Early Withdrawal | 57.5 (22.4) | 60.0 (23.3)
  SF-36v2 social function, Baseline | 76.1 (21.7) | 72.7 (28.3)
  SF-36v2 social function, Week 6 | 78.0 (21.4) | 77.6 (26.2)
  SF-36v2 social function, Week 14 | 73.4 (25.8) | 78.4 (22.6)
  SF-36v2 social function, Week 26/Early Withdrawal | 75.0 (25.8) | 79.0 (24.2)
  SF-36v2 emotional role, Baseline | 73.4 (25.4) | 69.1 (30.9)
  SF-36v2 emotional role, Week 6 | 73.1 (24.6) | 77.5 (25.9)
  SF-36v2 emotional role, Week 14 | 73.3 (22.9) | 74.1 (25.2)
  SF-36v2 emotional role, Week 26/Early Withdrawal | 71.5 (26.5) | 76.9 (25.4)
  SF-36v2 mental health, Baseline | 70.3 (18.7) | 68.0 (21.0)
  SF-36v2 mental health, Week 6 | 71.7 (18.3) | 71.8 (19.0)
  SF-36v2 mental health, Week 14 | 68.6 (20.4) | 70.6 (19.3)
  SF-36v2 mental health, Week 26/Early Withdrawal | 68.6 (22.8) | 70.2 (21.6)
  SF-36v physical component summary, Baseline | 45.6 (8.3) | 46.9 (9.7)
  SF-36v physical component summary, Week 6 | 46.2 (8.3) | 48.7 (9.0)
  SF-36v physical component summary, Week 14 | 46.3 (8.3) | 49.0 (8.1)
  SF-36v physical component summary, Week 26/EW | 46.2 (8.1) | 48.7 (8.6)
  SF-36v2 mental component summary, Baseline | 46.4 (10.1) | 44.3 (12.6)
  SF-36v2 mental component summary, Week 6 | 46.8 (10.0) | 47.2 (11.1)
  SF-36v2 mental component summary, Week 14 | 45.3 (11.1) | 46.2 (11.3)
  SF-36v2 mental component summary, Week 26/EW | 45.2 (12.3) | 46.5 (12.4)

8. Secondary Outcome: HR-QoL Instrument and Domain Scores From the FACIT-F Questionnaire at Baseline, Week 6, Week 14, and Week 26 or Early Discontinuation From Study Treatment
Description: Health-related quality of life (HR-QoL) patient reported outcomes from the functional assessment of chronic illness therapy fatigue (FACIT-F) questionnaire. Scores could range from 0 (worst possible) to 52 (best possible).
Time Frame: Baseline, Week 6, Week 14, and Week 26/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Points on a scale (0-52)
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Points on a scale (0-52)
  Baseline | 36.3 (9.0) | 36.0 (12.2)
  Week 6 | 38.3 (8.2) | 39.2 (9.7)
  Week 14 | 36.9 (10.2) | 39.5 (9.9)
  Week 26/Early Withdrawal | 37.0 (11.3) | 39.2 (10.1)

9. Secondary Outcome: HR-QoL Instrument and Domain Scores for the FACT-Th Questionnaire at Baseline, Week 6, Week 14, and Week 26 or Early Discontinuation From Study Treatment
Description: Health-related quality of life (HR-QoL) patient reported outcomes from the functional assessment of cancer therapy thrombocytopenia (FACT-Th) questionnaire (six selected items). Scores could range from 0 (worst possible) to 24 (best possible).
Time Frame: Baseline, Week 6, Week 14, and Week 26/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Points on a scale (0-24)
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Points on a scale (0-24)
  Baseline | 14.8 (5.8) | 13.5 (5.8)
  Week 6 | 15.1 (5.7) | 15.9 (6.0)
  Week 14 | 15.3 (5.4) | 16.7 (5.6)
  Week 26/Early Withdrawal | 15.3 (6.0) | 16.0 (6.1)

10. Secondary Outcome: HR-QoL Instrument and Domain Scores From the MEI-SF Questionnaire at Baseline, Week 6, Week 14, and Week 26 or Early Discontinuation From Study Treatment
Description: Health-related quality of life (HR-QoL) patient reported outcomes from the motivation and energy inventory-short form (MEI-SF) questionnaire. Scores could range from 0 (worst possible) to 72 (best possible).
Time Frame: Baseline, Week 6, Week 14, and Week 26/Early Withdrawal
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Points on a scale (0-72)
Arm/Group | Placebo | Eltrombopag 50 mg QD
Number analyzed (Participants) | 62 | 135
Points on a scale (0-72)
  Baseline | 71.3 (17.2) | 72.7 (21.4)
  Week 6 | 73.4 (16.4) | 76.2 (19.5)
  Week 14 | 71.1 (20.5) | 76.9 (20.5)
  Week 26/Early Withdrawal | 72.0 (21.7) | 76.7 (20.2)

ADVERSE EVENTS:
Description: 62 participants were randomized to the placebo arm, but only 61 took study medication and are analyzed in the Safety Population.
Arm/Group | Placebo | Eltrombopag 50 mg QD
Serious Adverse Events (participants affected / at risk) | 11/61 | 16/135
Other Adverse Events (participants affected / at risk) | 56/61 | 120/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | Eltrombopag 50 mg QD (N=135)
Cataract (Eye disorders) | 2 | 2
Cataract subcapsular (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 3
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Alanine aminotransferase (ALT) increased (Investigations) | 1 | 1
Aspartate aminotransferase (AST) increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Renal function test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=61) | Eltrombopag 50 mg QD (N=135)
Nasopharyngitis (Infections and infestations) | 12 | 14
Upper respiratory tract infection (Infections and infestations) | 7 | 14
Urinary tract infection (Infections and infestations) | 4 | 8
Influenza (Infections and infestations) | 3 | 7
Pharyngitis (Infections and infestations) | 1 | 9
Cellulitis (Infections and infestations) | 4 | 1
Headache (Nervous system disorders) | 20 | 40
Dizziness (Nervous system disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 17
Nausea (Gastrointestinal disorders) | 4 | 17
Abdominal pain upper (Gastrointestinal disorders) | 5 | 7
Constipation (Gastrointestinal disorders) | 6 | 6
Vomiting (Gastrointestinal disorders) | 1 | 10
Dyspepsia (Gastrointestinal disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Conjunctival haemorrhage (Eye disorders) | 3 | 3
Fatigue (General disorders) | 8 | 13
Oedema peripheral (General disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Alanine aminotransferase (ALT) increased (Investigations) | 3 | 9
Aspartate aminotransferase (AST) increased (Investigations) | 2 | 7
Insomnia (Psychiatric disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.